CLINICAL TRIAL: NCT01348542
Title: Efficacy of Trazodone vs. Cognitive Behavioral Therapy in Patients With Chronic Insomnia Associated With Objective Short Sleep Duration
Brief Title: Study of Trazodone & Cognitive Behavioral Therapy to Treat Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Alexandros Vgontzas, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35933
Record Dates: First submitted 2011-04-20; First posted 2011-05-05 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Insomnia
Keywords: Chronic Insomnia; Short Sleep Duration; Trazodone; Cognitive Behavioral Therapy; Efficacy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Trazodone; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trazodone (Active Comparator)
  Interventions: Drug: Trazodone
- Cognitive Behavioral Therapy (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Trazodone — 50 mg once a day, for 3 months
  Arms: Trazodone
Behavioral: Cognitive Behavioral Therapy — The CBT Protocol is implemented over a period of 12 weeks, with 4 consultations held on a weekly basis and 4 held on a biweekly basis.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to evaluate the effect of a 3 month medication trial of Trazodone versus 3 months of Cognitive Behavioral Therapy (CBT) in patients with chronic insomnia.

DETAILED DESCRIPTION:
Participants with chronic insomnia associated with objective short sleep duration will be recruited to participate in a 3 month clinical trial on the efficacy of trazodone versus CBT, with a 6 month follow up. The primary outcome measure will be objective sleep duration as measured by both actigraphy and polysomnography. The secondary outcome measure will be subjective severity of sleep disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic insomnia with duration of more than 1 year
* Objective short sleep duration (< 6 hours)
* BMI < 39
* Ages 30-60
* Men & Women

Exclusion Criteria:

* Major Mental Illness
* Substance Abuse/Dependence
* Sleep Apnea
* Periodic Limb Movement Disorder
* Shift Work or circadian disorders
* Diabetes
* Chronic Renal Failure, Hepatic Insufficiency, Chronic Heart Failure
* Current Use of hypnotics or sleep inducing sedative antidepressants

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros N Vgontzas, MD, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Vgontzas AN, Liao D, Pejovic S, Calhoun S, Karataraki M, Basta M, Fernandez-Mendoza J, Bixler EO. Insomnia with short sleep duration and mortality: the Penn State cohort. Sleep. 2010 Sep;33(9):1159-64. doi: 10.1093/sleep/33.9.1159. PMID 20857861
- [Background] Vgontzas AN, Liao D, Pejovic S, Calhoun S, Karataraki M, Bixler EO. Insomnia with objective short sleep duration is associated with type 2 diabetes: A population-based study. Diabetes Care. 2009 Nov;32(11):1980-5. doi: 10.2337/dc09-0284. Epub 2009 Jul 29. PMID 19641160
- [Background] Vgontzas AN, Liao D, Bixler EO, Chrousos GP, Vela-Bueno A. Insomnia with objective short sleep duration is associated with a high risk for hypertension. Sleep. 2009 Apr;32(4):491-7. doi: 10.1093/sleep/32.4.491. PMID 19413143
- [Background] Vgontzas AN, Bixler EO, Lin HM, Prolo P, Mastorakos G, Vela-Bueno A, Kales A, Chrousos GP. Chronic insomnia is associated with nyctohemeral activation of the hypothalamic-pituitary-adrenal axis: clinical implications. J Clin Endocrinol Metab. 2001 Aug;86(8):3787-94. doi: 10.1210/jcem.86.8.7778. PMID 11502812
- [Background] Fernandez-Mendoza J, Calhoun S, Bixler EO, Pejovic S, Karataraki M, Liao D, Vela-Bueno A, Ramos-Platon MJ, Sauder KA, Vgontzas AN. Insomnia with objective short sleep duration is associated with deficits in neuropsychological performance: a general population study. Sleep. 2010 Apr;33(4):459-65. doi: 10.1093/sleep/33.4.459. PMID 20394314
- [Background] Fernandez-Mendoza J, Calhoun SL, Bixler EO, Karataraki M, Liao D, Vela-Bueno A, Jose Ramos-Platon M, Sauder KA, Basta M, Vgontzas AN. Sleep misperception and chronic insomnia in the general population: role of objective sleep duration and psychological profiles. Psychosom Med. 2011 Jan;73(1):88-97. doi: 10.1097/PSY.0b013e3181fe365a. Epub 2010 Oct 26. PMID 20978224
- [Derived] Li Y, Vgontzas AN, Fernandez-Mendoza J, Fang J, Puzino K, Bixler EO. Effect of trazodone versus cognitive-behavioural treatment on high- and slow-frequency activity during non-rapid eye movement sleep in chronic insomnia: A pilot, randomized clinical trial. J Sleep Res. 2021 Oct;30(5):e13324. doi: 10.1111/jsr.13324. Epub 2021 Mar 5. PMID 33675113
- [Derived] Vgontzas AN, Puzino K, Fernandez-Mendoza J, Krishnamurthy VB, Basta M, Bixler EO. Effects of trazodone versus cognitive behavioral therapy in the insomnia with short sleep duration phenotype: a preliminary study. J Clin Sleep Med. 2020 Dec 15;16(12):2009-2019. doi: 10.5664/jcsm.8740. PMID 32780015

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trazodone | Cognitive Behavioral Therapy
Started | 13 | 11
Completed | 10 | 11
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trazodone | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (8.75) | 45.27 (9.94) | 44.0 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 9 | 18
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 11 | 21
Insomnia Severity Index [Mean (Standard Deviation); unit: score on a scale] — The Insomnia Severity Index (ISI) a self completed questionnaire was used to measure the severity of sleep disturbance. The ISI is composed of 7 items each rated on a scale of 0-4. The total score was calculated by adding the individual item scores. The total ISI Scale can range from 0-28 with higher total scores indicating a higher severity of insomnia symptoms and sleep disturbance.
  score on a scale | 16.70 (3.59) | 16.18 (2.18) | 16.43 (2.87)

OUTCOME MEASURES:

1. Primary Outcome: Change in Objective Polysomnography Sleep Duration From Baseline to Post Treatment (3 Months)
Description: Polysomnography (8 hours fixed time in bed) will be used to measure sleep duration at baseline and post treatment (3 months)
Time Frame: Baseline to Post Treatment (3 months)
Population: Objective Short Sleepers defined by 2 week actigraphy sleep duration measurement
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Trazodone | Cognitive Behavioral Therapy
Number analyzed (Participants) | 7 | 8
minutes | 28.95 (31.70) | 38.91 (24.74)

2. Primary Outcome: Change in Objective Polysomnography Sleep Duration From Baseline to Follow up (9 Months)
Description: Polysomnography (8 hours fixed time in bed) will be used to measure sleep duration at baseline and follow up (9 months)
Time Frame: Baseline to follow up (9 months)
Population: From the 21 participants who completed the study, 15 met the criteria for objective short sleep duration and were included in the final analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Trazodone | Cognitive Behavioral Therapy
Number analyzed (Participants) | 7 | 8
minutes | 51.78 (76.39) | 32.36 (30.31)

3. Primary Outcome: Change in Objective Actigraphy Sleep Duration From Baseline to Post Treatment (3 Months)
Description: Actigraphy (ad libitum time in bed) will be used to measure sleep duration at baseline and Post Treatment (3 months)
Time Frame: Baseline to Post Treatment (3 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Trazodone | Cognitive Behavioral Therapy
Number analyzed (Participants) | 7 | 8
minutes | 51.01 (57.50) | -11.73 (31.43)

4. Primary Outcome: Change in Objective Actigraphy Sleep Duration From Baseline to Follow up (9 Months)
Description: Actigraphy (ad libitum time in bed) will be used to measure sleep duration at baseline and follow up (9 months)
Time Frame: Baseline to follow up (9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Trazodone | Cognitive Behavioral Therapy
Number analyzed (Participants) | 7 | 8
minutes | 50.35 (27.47) | -7.56 (38.04)

5. Secondary Outcome: Change From Baseline in Subjective Severity of Sleep Disturbance at 3 Months
Description: The Insomnia Severity Index (ISI) was used to measure the change in severity of sleep disturbance at baseline to post treatment (3 months). The ISI is composed of 7 items each rated on a scale of 0-4. The total score was calculated by adding the individual item scores. The total ISI scale score ranged from 0-28 with higher total scores indicating a higher severity of insomnia symptoms.
Time Frame: Baseline to Post Treatment (3 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trazodone | Cognitive Behavioral Therapy
Number analyzed (Participants) | 7 | 8
score on a scale | -12.29 (4.35) | -10.75 (2.87)

6. Secondary Outcome: Change From Baseline in Subjective Severity of Sleep Disturbance at 9 Months
Description: The Insomnia Severity Index (ISI) was used to measure the change in severity of sleep disturbance at baseline to Follow Up (9 months). The ISI is composed of 7 items each rated on a scale of 0-4. The total score was calculated by adding the individual item scores. The total ISI scale score ranged from 0-28 with higher total scores indicating a higher severity of insomnia symptoms.
Time Frame: Baseline to follow up (9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trazodone | Cognitive Behavioral Therapy
Number analyzed (Participants) | 7 | 8
score on a scale | -13.29 (3.77) | -10.38 (3.02)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Trazodone | Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT01348542/Prot_SAP_000.pdf